CLINICAL TRIAL: NCT06913985
Title: Trajectory Study: Predicting Cardiometabolic Health in Adolescents and Young Adults Based on Childhood Fitness, Sleep, and Diet
Acronym: Trajectory
Status: Enrolling by invitation | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 297969
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-05

CONDITIONS: Cardiometabolic Health
Keywords: diet; physical fitness; adolescents; children; longitudinal study; diet quality; sleep quality; cardiovascular risk prediction
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Trajectory study aims to determine whether childhood aerobic fitness, sleep quality, and diet quality predict cardiometabolic health during puberty and early adulthood, independently of adiposity.

DETAILED DESCRIPTION:
The Trajectory study is a longitudinal observational study. Participants will be recalled from two existing pediatric cohorts: the Arkansas Active Kids study (ClinicalTrials.gov ID: NCT03221673; IRB #206217) and the MI Energy study (ClinicalTrials.gov ID: NCT04427462; IRB #260376). Both were cross-sectional studies with comparable designs, recruiting children between ages 7 and 10 years, regardless of sex, BMI, or ethnicity. The Trajectory study serves as the follow-up component during adolescence or early adulthood (ages 13-21). It is anticipated that approximately 250 participants will complete the follow-up visit.

During the follow-up visit at the Arkansas Children's Nutrition Center (ACNC), the following key measurements will be conducted:

* Body Composition: Dual-Energy X-ray Absorptiometry (DXA)
* Metabolic Profile: Fasting blood markers, including glucose, lipid profile, and insulin resistance
* Continuous Glucose Monitoring: Interstitial sensor-based glucose
* Vascular Function: Ultrasound (brachial artery flow-mediated dilation)
* Liver Examination: Ultrasound (liver steatosis and stiffness)
* Resting Metabolic Rate: Indirect calorimetry
* Aerobic Capacity: Cardiopulmonary exercise test (spirometry)
* Muscle Strength: Dynamometry
* Physical Activity & Sleep: Accelerometry
* Dietary Intake: Food frequency questionary

ELIGIBILITY:
Inclusion Criteria:

* Ages 13 to 21 years.
* Boys or girls.
* All ethnicities.
* All BMIs.
* Previous participation in the Arkansas Active Kids study and the MI Energy study.
* Participants who previously agreed to be contacted for future research at ACNC.
* Participants who agree to the use of their previously collected information and samples from the AAK or MI Energy studies for the follow-up study.

Exclusion Criteria:

* Asthma that requires daily use of inhalers to keep symptoms under control.
* Asthma that requires use of rescue inhalers (e.g., albuterol) >2 days per week.
* Exercise-induced asthma.
* Autism spectrum disorder (e.g., Autistic disorder, Rett disorder, Asperger disorder, childhood disintegrative disorder, pervasive developmental disorder not otherwise specified (PDD-NOS).
* Neurological disorders (e.g. epilepsy or seizures).
* Cancer.
* Hormonal disease (e.g., hypothyroidism and growth hormone deficiency).
* Autoimmune diseases (e.g., lupus, thyroiditis, juvenile idiopathic arthritis).
* Bleeding disorders (e.g., hemophilia).
* Chronic infections (e.g., HIV, hepatitis B, hepatitis C).
* Other pre-existing medical conditions or medications as determined by the investigators to affect the outcomes of interest.
* Pregnancy (verbal assessment).

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents (13 to 17 years) and young adults (18 to 21 years) who previously participated in the Arkansas Active Kids study (clinicaltrials.gov #NCT03221673; IRB #206217) and the MI Energy study (clinicaltrials.gov #NCT04427462; IRB #260376).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite score of cardiometabolic health status. | Baseline assessment in childhood (ages 7-10) and follow-up assessment during adolescence or early adulthood (ages 13-21)
  This composite outcome evaluates cardiometabolic health across two time points (pre-/early-adolescence and adolescence/early adulthood). It is calculated as the mean of z-scores for: fasting triglycerides and total cholesterol/HDL ratio (from fasting blood samples), HOMA2-IR (from fasting glucose and insulin), systolic blood pressure (automated sphygmomanometer), fat mass index [DXA-derived fat mass (kg)/height²], and inverse peak oxygen uptake (measured via graded exercise test with indirect calorimetry). The composite provides an overall measure of cardiometabolic health status. The goal is to assess whether childhood aerobic fitness, sleep quality, and diet quality independently predict this score, controlling for adiposity [DXA-derived fat mass index (kg/m²)].

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Borsheim, Ph.D, Principal Investigator — Arkansas Children's Research Institute
Locations (2):
- United States (2):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Arkansas Children's Nutrition Center, Little Rock, Arkansas

IPD SHARING:
Plan to Share IPD: Undecided